CLINICAL TRIAL: NCT01993914
Title: Prevalence of MTHFR Polymorphisms in Venous Disease With or Without Concomitant Thrombosis
Brief Title: Prevalence of MTHFR Polymorphisms in Venous Disease
Acronym: MTHFR
Status: Completed | Type: Observational
Sponsor: Health Diagnostic Laboratory, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R2011-2104
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Varicose Veins; MTHFR; Venous Disease; Thrombosis
MeSH Terms: conditions — Varicose Veins; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood and serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The etiologies of varicose veins and the progression to more serious forms of chronic venous disease and identification of appropriate diagnostic tests to better aid patient management by identifying individuals who may benefit from more aggressive treatment and/ or prophylactic measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* No venous disease (N=30); or C2-C3 venous disease (N=30); or C4-C6 venous disease (N=30)

Exclusion Criteria:

* Pregnancy
* Cancer
* Chronic obstructive pulmonary disease (COPD)
* Any systemic inflammatory disease
* Any of the following within the previous 30 days:

  * Trauma
  * Any surgery
  * Periods of prolonged inactivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the Elite Laser Vein Center, representative of the ethnic population of Los Angeles, CA, estimated as 40% Non Hispanic White, 40% Hispanic, 10% African American, 10% Asian.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of MTHFR mutation between patients | Baseline
  Determine whether the prevalence of the MTHFR mutation differs between patient with varicose veins compared to controls and with or without superficial vein thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Richman, MD,FACS,FCCP, Principal Investigator
Locations (1):
- The Elite Laser Vein Center, Los Angeles, California, United States

REFERENCES:
- [Background] Sverdlova AM, Bubnova NA, Baranovskaya SS, Vasina VI, Avitisjan AO, Schwartz EI. Prevalence of the methylenetetrahydrofolate reductase (MTHFR) C677T mutation in patients with varicose veins of lower limbs. Mol Genet Metab. 1998 Jan;63(1):35-6. doi: 10.1006/mgme.1997.2638. No abstract available. PMID 9538515
- [Background] Wilmanns C, Casey A, Schinzel H, Walter PK. Superficial thrombophlebitis in varicose vein disease: the particular role of methylenetetrahydrofolate reductase. Phlebology. 2011 Jun;26(4):135-9. doi: 10.1258/phleb.2009.009075. Epub 2010 Sep 29. PMID 20881312
- [Background] Krijnen RM, de Boer EM, Bruynzeel DP. Epidemiology of venous disorders in the general and occupational populations. Epidemiol Rev. 1997;19(2):294-309. doi: 10.1093/oxfordjournals.epirev.a017959. No abstract available. PMID 9494789
- [Background] Campbell B. Varicose veins and their management. BMJ. 2006 Aug 5;333(7562):287-92. doi: 10.1136/bmj.333.7562.287. No abstract available. PMID 16888305
- [Background] Jorgensen JO, Hanel KC, Morgan AM, Hunt JM. The incidence of deep venous thrombosis in patients with superficial thrombophlebitis of the lower limbs. J Vasc Surg. 1993 Jul;18(1):70-3. doi: 10.1067/mva.1993.42072. PMID 8326661
- [Background] Ascer E, Lorensen E, Pollina RM, Gennaro M. Preliminary results of a nonoperative approach to saphenofemoral junction thrombophlebitis. J Vasc Surg. 1995 Nov;22(5):616-21. doi: 10.1016/s0741-5214(95)70049-8. PMID 7494365
- [Background] Chengelis DL, Bendick PJ, Glover JL, Brown OW, Ranval TJ. Progression of superficial venous thrombosis to deep vein thrombosis. J Vasc Surg. 1996 Nov;24(5):745-9. doi: 10.1016/s0741-5214(96)70007-1. PMID 8918318
- [Background] Leon L, Giannoukas AD, Dodd D, Chan P, Labropoulos N. Clinical significance of superficial vein thrombosis. Eur J Vasc Endovasc Surg. 2005 Jan;29(1):10-7. doi: 10.1016/j.ejvs.2004.09.021. PMID 15570265
- [Background] Binder B, Lackner HK, Salmhofer W, Kroemer S, Custovic J, Hofmann-Wellenhof R. Association between superficial vein thrombosis and deep vein thrombosis of the lower extremities. Arch Dermatol. 2009 Jul;145(7):753-7. doi: 10.1001/archdermatol.2009.123. PMID 19620555
- [Background] Caprini JA, Goldshteyn S, Glase CJ, Hathaway K. Thrombophilia testing in patients with venous thrombosis. Eur J Vasc Endovasc Surg. 2005 Nov;30(5):550-5. doi: 10.1016/j.ejvs.2005.05.034. Epub 2005 Aug 1. PMID 16055356